CLINICAL TRIAL: NCT06550817
Title: Growth Mindset Intervention Improves Positive Response to E-Health for Older Adults With Chronic Disease: A Randomized Controlled Trial
Brief Title: Growth Mindset Intervention for Older Adults With Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huzhou University (Other)
Responsible Party: Principal Investigator, Yaling Zeng, Principal Investigator, Huzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022015
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- growth mindset + e-health (Experimental): Participants received an e-health program intervention plus a growth mindset intervention over 12 weeks, with weekly sessions for the first 6 weeks and biweekly follow-up phone calls for the next six weeks.
  Interventions: Other: Growth mindset intervention
- e-health only (Active Comparator): Participants received an e-health program intervention over 12 weeks, with weekly sessions for the first 6 weeks and biweekly follow-up phone calls for the next six weeks.
  Interventions: Other: E-health Program

INTERVENTIONS:
Other: Growth mindset intervention — Online intervention is implemented and it lasts about 20 minutes each time, while face-to-face intervention lasts about 30 minutes each time, and they are carried out for a total of six weeks, face-to-face or telephone intervention is implemented once every two weeks for about 15 minutes each time
  Arms: growth mindset + e-health
Other: E-health Program — face-to-face e-health teaching in the first 6 weeks, and telephone follow-up were conducted once a week, for about 10 minutes each time in the last 6 weeks
  Arms: e-health only

SUMMARY:
This study was conducted to develop and investigate the effectiveness of a growth mindset intervention based on growth mindset theory.

DETAILED DESCRIPTION:
The study employed a quasi-randomized controlled trial design conducted over 12 weeks. Before conducting the study, the researchers numbered the wards of internal medicine departments (excluding intensive care units) according to the order of bed number. The wards were then randomly divided into intervention wards and control wards using a random number generator. Patients were recruited to the control group (e-health only) in the control ward and the intervention group (growth mindset intervention+ e-health) in the intervention unit. Participants in the control group could undergo the training after the study concluded.

ELIGIBILITY:
Inclusion Criteria:

* aged≥60 years
* diagnosed≥1 chronic disease
* owned at least one smartphone
* could communicate clearly in writing or orally
* were willing to participate in this study

Exclusion Criteria:

* could not use WeChat or phone to communicate
* diagnosed as mental illness or cognitive impairment
* suffered from acute severe disease or lost self-care ability
* undergoing other similar training

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Implicit Theories of Intelligence Scale-6 | Baseline,Week 6, and Week 12
  The Implicit Theories of Intelligence Scale-6 (ITIS-6) is a validated, self-reported instrument assessing participants' level of growth mindset. A mean score of greater than or equal to 4 on all items indicates that the individual has a growth mindset, and vice versa for a fixed mindset.
Questionnaire of Knowledge, Willingness, Confidence, and Practice of Smart Medicine (KWCP-SM) | Baseline,Week 6, and Week 12
  The Questionnaire of Knowledge, Willingness, Confidence, and Practice of Smart Medicine (KWCP-SM) is a validated, self-reported instrument assessing participants' level of knowledge, willingness, confidence, and practice of smart medicine. The questionnaire adopted the Likert-5 scoring method. The higher score indicated a higher level of knowledge, willingness, confidence, and practice of smart medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Meijuan Cao, Study Chair — Huzhou University
Locations (2):
- China (2):
  - School of Medicine and Nursing， Huzhou University, Huzhou, Zhejiang
  - School of Nursing Huzhou University, Huzhou, Zhejiang